CLINICAL TRIAL: NCT02629068
Title: Parents United With Responsive Parents for Online Support and Education PURPOSE: A Social Media Intervention for Parent Support
Brief Title: PURPOSE: A Social Media Intervention for Parent Support
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants were enrolled in the pilot phase of the study due to lack of interest from parents. Completion dates reflect the end of funding for the study.
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Marya Schulte, Clinical Psychologist, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21DA039459 (NIH); R21DA039459 (NIH)
Record Dates: First submitted 2015-11-30; First posted 2015-12-11 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Substance Use Disorders; Parenting
Keywords: Adolescent; Social Support; Social Media; Parents; Shame; Stigma
MeSH Terms: conditions — Substance-Related Disorders; Social Stigma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PURPOSE (Experimental): Parents in the PURPOSE group will join a "secret" Facebook group for 2 months. Groups will be lead by 2 peer leaders and include 20 parent participants.
  Interventions: Behavioral: PURPOSE
- Treatment as Usual (TAU) (No Intervention): Treatment as Usual parents will be contacted after 8 weeks to complete follow-up interview. Will not receive PURPOSE intervention.

INTERVENTIONS:
Behavioral: PURPOSE — The first week of the intervention will focus on welcoming everyone to the facebook group and laying down the ground rules for participation. Each additional week of the intervention will focus on a specific topic to promote discussion and learning of each particular skill; however, questions and discussions on other relevant topics are always welcome and encouraged.
  Week 1: Welcome Week Week 2: SUD Basics Week 3: Problem of Stigma Week 4: Communication Skills Week 5: Parental Monitoring Week 6: Stress Management Week 7: Family and Valued Directions Week 8: Putting It All Together
  Arms: PURPOSE

SUMMARY:
The purpose of this study is to develop and test a social media-based (Facebook) intervention that provides support and skills to parents with adolescent children in treatment for substance abuse. The Facebook intervention, PURPOSE, will be 8 weeks long and led by other parents (peer leaders). Peer leaders will go through 2 2-3-hour training sessions and be assessed at the end to confirm their understanding of study protocol and procedures. The study PI will lead 2 short (2-weeks) trial tests of various segments of the intervention to test out content and procedures. Then, a pilot trial with 80 parents, 40 randomized to PURPOSE and 40 randomized to treatment as usual (TAU), will be done to test how useful PURPOSE can be in promoting parents' engagement in their child's treatment and recovery while reducing their own distress and feelings of shame/stigma. Parents will do a phone interview at the start of PURPOSE and again at the end of the 8 weeks.

DETAILED DESCRIPTION:
This study will take advantage of established peer training techniques to train parents of adolescents who are more experienced to help other parents better engage in services for their adolescent child. This pilot study marks the beginning of our long-term program of research focused on adapting intervention tools for delivery via e-technology platforms as a means for optimizing treatment effectiveness for youth. Thus, the proposed study will contribute to the scientific literature on the role of parental support in adolescent recovery as well as respond to NIDA's call for increased understanding of the feasibility and utility of social media as an option expanding the traditional treatment and face-to-face self-help groups. The proposed study has the following aims:

Aim 1: To develop PURPOSE, a social-media based intervention that provides information and coping tools for parents/guardians of adolescent children with a SUD. The theoretically grounded intervention will be peer-led, and will be developed and refined with feedback from experts, providers, parents, and adolescents.

Aim 2: To determine the feasibility and acceptability of PURPOSE that uses online peer-led intervention delivery. Trial testing will be conducted to iteratively refine content and procedures in order to optimize the engagement and usefulness of the intervention for parents.

Aim 3: To conduct a pilot control trial to provide preliminary data on this intervention so as to determine if social media-based parent support group involvement positively impacts parent outcomes (reduced stigma and distress, improved parent monitoring, and increased engagement in adolescent treatment) and adolescent outcomes (treatment retention and abstinence).

ELIGIBILITY:
Inclusion Criteria:

* Be the parent/guardian of an adolescent (under age 18) currently receiving out-patient treatment for SUD
* Have an active Facebook and email account
* Be able to read and write English

Exclusion Criteria:

* Any medical and/or psychiatric conditions which would require immediate or ongoing treatment that would make study participation difficult or harmful
* Already participating in an online support group for parents of teens in treatment

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Adolescent Treatment History and Parental Engagement Questionnaire | 8 weeks
  Parental report of child's treatment status, including enrollment date, primary reason for seeking treatment, and type of facility. All parents will also report on number of informal parent/family support groups (e.g., AlAnon) and formal treatment sessions they have attended (baseline and follow-up).

SECONDARY OUTCOMES:
Perceived Stigma of Addiction Scale | 8 weeks
  The PSAS is an 8-item self-report questionnaire designed to assess perceptions of the prevalence of stigmatizing beliefs towards individuals with substance use diagnoses and treatment histories (baseline and follow-up)
Parental Monitoring Questionnaire | 8 weeks
  Relationship and disclosure constructs will be used from Stattin and Kerr's (2000) questionnaire of parental monitoring (baseline and follow-up)
Satisfaction and Usability Questionnaire | 8 weeks
  Participants will report overall satisfaction and degree to which information provided was deemed applicable and helpful. Likert-scale reports of satisfaction as well as responses to open-ended questions will be collected (PURPOSE intervention parents only and follow-up only).
K-10 Scale of Psychological Distress | 8 weeks
  The U.S. National Health Survey K-10 is a 10-item screening scale used to assess the degree of non-specific psychological distress over the past 30 days (baseline and follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: Marya Schulte, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Integrated Substance Abuse Programs, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No